CLINICAL TRIAL: NCT07032233
Title: Assessment of Lower Extremity Muscle Strength, Balance, and Functional Capacity in Individuals With Transfemoral Amputation and Investigation of the Relationship With the Length of the Lost Extremity
Brief Title: Assessment of Strength, Balance, and Function in Above-Knee Amputees in Relation to Residual Limb Length
Status: Not yet recruiting | Type: Observational
Sponsor: Ceren Kuzu (Other)
Collaborators: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other); Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Ceren Kuzu, PhD Candidate, Physiotherapist, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: FTREK25/31
Record Dates: First submitted 2025-06-06; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Transfemoral Amputation
Keywords: Transfemoral Amputation; Muscle Strength; Isokinetic Dynamometry; Balance Assessment; Functional Capacity; Residual Limb Length; Prosthetics; Postural Control; Gait; Six-Minute Walk Test; Mobility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- transfemoral amputation: Adults with unilateral transfemoral amputation who indepently ambulates with a prosthetic limb.

SUMMARY:
The goal of this observational study is to learn how muscle strength, balance, and functional ability are affected in people with above-knee (transfemoral) amputations. The main questions it aims to answer are:

How does the length of the lost part of the leg, compared to the intact leg, affect muscle strength, balance, and functional capacity?

Is muscle strength at specific lower limb joints related to balance and performance ?

Participants will:

Have muscle strength measured at all intact lower limb joints using an isokinetic dynamometer

Complete balance assessments using force platform technology that measures weight distribution and evaluates both static and dynamic balance

Perform a six-minute walk test to evaluate endurance and functional capacity

The study will help improve understanding of how limb length and joint-specific muscle strength impact mobility, supporting the development of better rehabilitation programs for amputees.

DETAILED DESCRIPTION:
This study is a cross-sectional observational study designed to assess lower extremity muscle strength, balance, and functional capacity in individuals with unilateral transfemoral amputation. The primary aim is to examine how the length of the lost part of the limb, in relation to the intact limb, correlates with these physical performance parameters. This study does not involve any intervention or follow-up over time. All data will be collected at one time point. Therefore, although the registry requires a study model selection, the study design does not align with standard cohort or case-control models. For this reason, the "Other" option was selected as the most appropriate observational study model.

ELIGIBILITY:
Inclusion Criteria:

Individuals will be included in the study if they:

Are between 18 and 50 years of age

Are literate

Have unilateral transfemoral amputation

Have no cardiovascular, orthopedic, cognitive, or neurological conditions that could negatively affect balance, gait, or muscle strength

Are able to ambulate independently with a prosthesis

Have been walking for at least 6 months

Voluntarily agree to participate in the study

Exclusion Criteria:

Participants will be excluded from the study if:

They develop complications such as pain (rated 3 or higher on the Visual Analog Scale) or stump irritation during the course of the study

Their residual limb length is less than 25 cm from the greater trochanter, which exceeds the limitations of the isokinetic dynamometer attachments used in the study

They voluntarily withdraw from the study - in such cases, their data will be removed from the records

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be selected from the population of adults with unilateral transfemoral amputation who are able to ambulate independently with a prosthesis. The target population includes individuals between the ages of 18 and 50 who have been using a prosthesis for at least 6 months. Eligible participants must be literate and free from cardiovascular, orthopedic, cognitive, or neurological conditions that could interfere with gait, balance, or muscle strength. Recruitment may occur through rehabilitation clinics, prosthetics centers, or community referrals.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Length of Residual Limb and Intact Limb (cm) and Percentage of Limb Loss (%) | 1 day
  Anthropometric measurements will be performed using a standard measuring tape. For the amputated limb, the distance will be measured from the greater trochanter to the distal end of the residual limb along the lateral midline. For the intact limb, the measurement will extend from the greater trochanter to the plantar surface of the foot. The difference between these two measurements will represent the length of the lost limb. The percentage of limb loss will then be calculated by comparing the lost length to the total length of the intact limb.
Isokinetic Strength Testing | 5 days
  Isokinetic muscle strength assessments will be conducted using the IsoMed 2000 Dynamometer (D&R Ferstl GmbH, Hemau, Germany). Measurements will include peak torque (Nm) and total work (J) values for hip, knee, and ankle flexor/extensor muscles. Testing will be performed under the following angular velocities and repetitions:
  1. Hip Flexion/Extension: 5 reps at 60°/s, 10 reps at 120°/s (supine position)
  2. Knee Flexion/Extension: 5 reps at 60°/s, 10 reps at 180°/s (seated, hip at 90°)
  3. Ankle Plantar/Dorsiflexion: 5 reps at 60°/s, 10 reps at 120°/s (seated, semi-flexed hip, 90° knee flexion) Rest periods will be given between measurements to minimize fatigue. Tests will be randomized across different joints and days to avoid order effects.
  Data will be summarized as peak torque and total work values for each muscle group at the specified angular velocities.
Stability Coefficient (Eyes Open and Closed), Single-Leg Stability of Intact Side, and Limits of Stability (mm) | 1 day
  Participants' balance abilities will be assessed using the Huber 360® Evolution (LPG Systems, Valence, France), a motorized multi-axial platform with integrated force sensors. The following parameters will be measured and reported:
  1. Static balance with eyes open and eyes closed (coefficient of stability)
  2. Single-Leg Stability on the intact limb (coefficient of stability)
  3. Limits of stability quantified as sway in mm
6 minute walk test | 1 day

SECONDARY OUTCOMES:
The Amputee Mobility Predictor (AMP) | 1 day
  Mobility level will be assessed using the Amputee Mobility Predictor (AMP) scale. This performance-based tool includes 21 items covering balance while sitting, transfers, standing balance, walking, stair climbing, and assistive device use. Scores range from 0 to 47, with higher scores indicating better mobility. Based on the scores, participants will be classified according to the Medicare Functional Classification Levels (K-levels), which are defined by the United States Centers for Medicare & Medicaid Services (CMS) to standardize functional mobility and prosthetic eligibility.
The Comprehensive Lower-limb Amputee Socket Survey (CLASS) | 1 day
  Socket fit and comfort will be evaluated using The Comprehensive Lower-limb Amputee Socket Survey (CLASS), a validated self-report questionnaire developed by Gailey et al. The survey includes 15 items assessing four domains: stability, suspension, comfort, and appearance of the prosthetic socket. Each item is rated on a 4-point ordinal scale, and total scores are converted into a percentage score ranging from 0% to 100%, with higher percentages indicating better socket fit and greater user satisfaction.

OTHER OUTCOMES:
Information regarding amputation history and prosthesis use and demographics | 1 day

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, it is undecided whether individual participant data (IPD) will be shared. This study is part of an early-stage academic research project, and decisions regarding data sharing will depend on institutional policies, data protection considerations, and future collaboration opportunities. If a data-sharing plan is established, the study record will be updated accordingly.